CLINICAL TRIAL: NCT00782808
Title: Peripheral Reservoir of HIV DNA in Monocytes Pivotal to Cognition in HIV
Status: Completed | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Assoc.Prof.Jintanat Ananworanich, M.D., Assoc.Prof, SEARCH Research Foundation
Other Study IDs: SEARCH 011
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
Keywords: HIV DNA in Monocytes
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 HIV DNA will be stratified by high
- 2 HIV DNA will be stratified by low

SUMMARY:
Sixty HIV participants will be enrolled and stratified by PBMC HIV DNA levels, either high (greater than or equal to 5000 copies/106 cells) or low (less than 5000 copies/106 cells). Individuals will be enrolled into each group until filled. Screening PBMC HIV DNA levels will be performed at SEARCH in real-time with less than one-week turn around time. All individuals will intend to initiate ARV due to meeting MOPH guidelines for such. The protocol team will work with the primary care physician to facilitate initiation of standard ARV care; however, initiation of ARV is not a requirement of the study and ARV will not be provided by the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individuals meeting MOPH criteria to initiate HAART and planning to initiate HAART within a month of screening.
* Consequently, all participants will have plasma CD4 counts at less than 250 cells.

Exclusion Criteria:

* Head injury with loss of consciousness greater than 1 hour or cognitive sequela
* Current/past illicit drug use or positive drug screen for methamphetamines, amphetamines, or cocaine at screening or entry.
* Any of the following laboratory abnormalities:

  * PT/PTT > the upper limit of normal (ULN) or INR > 1.1
  * Hemoglobin < 9.0 mg/dL
  * ALT > 5x ULN
  * serum creatinine > 2x ULN or creatinine clearance < 30 cc per min by Cockroft-Gault formula
* Acute illness within 30 days prior, persistent and active AIDS-defining OI of any organ system or autoimmune disease.
* Current or recent fevers or meningeal signs suggestive of CNS opportunistic infection
* CNS opportunistic infection, past or present (Patients diagnosed with opportunistic infection after CSF examination will be excluded from further analysis. In such a situation, an additional patient will be enrolled)
* History of pre-existing neurologic disease to include stroke, multiple sclerosis or psychiatric illness including schizophrenia, bipolar disorder, anxiety disorder, panic attacks, major depression, or post traumatic stress disorder. Patients with past depression that is controlled and patients with or minor depressive symptoms will be allowed to enroll.
* Known learning disability including dyslexia or unable to read or write basic Thai
* Positive Hepatitis C serology (Hepatitis C Ab)
* Confusion or other signs and symptoms of metabolic encephalopathy or delirium
* Other conditions that could explain neurocognitive decline in the opinion of the investigator such as hypothyroidism, vitamin B12 deficiency or neurosyphilis
* Pregnancy or metal objects that would preclude MRI

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected individuals meeting MOPH criteria to initiate HAART and planning to initiate HAART within a month of screening. Consequently, all participants will have plasma CD4 counts at less than 250 cells.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To determine the long-term relationship between cognition and HIV DNA in circulating PBMCs and monocytes (CD14+ PBMCs) among patients initiating HAART for the first time | After March 30, 2016

CONTACTS AND LOCATIONS:
Overall Officials: Victor Valcour, MD, Principal Investigator — University of Hawii
Locations (1):
- SEARCH Thailand, Bangkok, Thailand

REFERENCES:
- [Derived] Corley MJ, Sacdalan C, Pang APS, Chomchey N, Ratnaratorn N, Valcour V, Kroon E, Cho KS, Belden AC, Colby D, Robb M, Hsu D, Spudich S, Paul R, Vasan S, Ndhlovu LC; SEARCH010/RV254 and SEARCH013/RV304 study groups. Abrupt and altered cell-type specific DNA methylation profiles in blood during acute HIV infection persists despite prompt initiation of ART. PLoS Pathog. 2021 Aug 13;17(8):e1009785. doi: 10.1371/journal.ppat.1009785. eCollection 2021 Aug. PMID 34388205
- See also: South East Asia Research Collaboration with Hawaii — http://www.searchthailand.org